CLINICAL TRIAL: NCT04452747
Title: Artificial Induction of Labour in Full-term Singleton Pregnancy : Comparative Randomized Clinical Trial of Two Strategies (DINO-FIRST Versus BALLON-FIRST)
Brief Title: Artificial Induction of Labour in Full-term Singleton Pregnancy : Comparative Randomized Trial of Two Strategies
Acronym: BESTWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL19_0044; 7756 (Other: UH Montpellier)
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dino-first (Active Comparator): Labour will be induced by the use of the vaginal Dinoprostone system (Propess®) first.
  Interventions: Procedure: Vaginal Dinoprostone system (Propess®)
- Balloon-first (Active Comparator): Labour will be induced by the use of a cervix dilatation balloon first.
  Interventions: Procedure: Dilatation balloon

INTERVENTIONS:
Procedure: Vaginal Dinoprostone system (Propess®) — Labour will be induced using the vaginal Dinoprostone system (Propess®) as a first strategy
  Arms: Dino-first
Procedure: Dilatation balloon — Labour will be induced using a cervix dilatation balloon as a first strategy
  Arms: Balloon-first

SUMMARY:
Labour induction is an obstetrical procedure, which artificially starts the process of cervix dilation, in order to induce labour. Several methods of labour induction exist : mechanical ones (using dilatation balloons) or pharmacological ones (using prostaglandins or oxytocin). This trial aims to compare, in case of non-favourable cervix, the strategy of labour induction using the Propess® method first (Dino-first) versus the strategy beginning with the use of a dilatation balloon (Ballon-first), with respect of the usual practice and the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy
* Fetus with cephalic presentation
* Intact membranes between 37 and 42 weeks of amenorrhea
* Medical indication for labour induction according to the "Haute Autorité de Santé" (HAS) guidelines
* Unfavourable cervix (Bishop scoring < 7)
* Age > 18 years-old
* Person affiliated to a healthcare system
* Good understanding of the French language

Exclusion Criteria:

* Previous C-section or uterine incision
* Placenta previa
* Metrorrhagia of unknown origin
* Lethal foetal abnormality
* Hyperreactivity to one of the molecules used for the induction (dinoprostone or oxytocin) or to latex
* Subject participants to another biomedical research
* Subject under legal guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of vaginal deliveries | On the day of the delivery
  Rate of vaginal deliveries (both spontaneous or instrumentally assisted)

SECONDARY OUTCOMES:
Rate of spontaneous vaginal deliveries | On the day of the delivery
  Number of spontaneous vaginal deliveries
Rate of instrumentally assisted vaginal deliveries, including the reason for the assistance | On the day of the delivery
  Number of instrumentally assisted vaginal deliveries, including the reason for the assistance
Rate of C-section including the reason for the C-section | On the day of the delivery
  Number of C-section including the reason for the C-section. The reasons for the C-section can be : a failure of dilatation at the first stage of the labour (between 0 and 10 cm), an absence of foetal descent at the second stage of labour, a foetal reason or a maternal reason)
Timeframe between the beginning of the induction and the beginning of the labour | On the day of the delivery
  Time elapsed between the beginning of the induction and the beginning of the labour
Cumulated rate of spontaneous vaginal deliveries | at 12 hours, 24 hours and 48 hours
  Cumulated number of spontaneous vaginal deliveries at 12 hours, 24 hours and 48 hours
Rate of labour induction failure | On the day of the delivery
  Rate of labour induction failure is measure by the number of C-sections carried out due to a latency phase (0-6cm), which lasted more than 24 hours, together with the administration of oxytocin for at least 12 to 18 hours after the membranes artifically broke.
Rate of secondary or tertiary use of Propess, Foley catheter of intra-veinous oxytocin | On the day of the delivery
  Number of secondary or tertiary use of Propess, Foley catheter of intra-veinous oxytocin
Rate of peridural anaesthesia during labour | On the day of the delivery
  Number of peridural anaesthesia during labour
Rate of uterine hyperstimulation without impact on the foetus | On the day of the delivery
  Uterine hyperstimulation is described as a number of contractions of 6 or more within 10 minutes, repeating at least twice). Foetal impact is defined as a slowing of the foetal heart rate.
Rate of uterine hyperstimulation with an impact on the foetus | On the day of the delivery
  Uterine hyperstimulation is described as a number of contractions of 6 or more within 10 minutes, repeating at least twice). Foetal impact is defined as a slowing of the foetal heart rate.
Rate of uterine hypertonia | On the day of the delivery
  Uterine hypertonia is describes as a frequency of contractions every 2 minutes or less together with a slowing of the foetal heart rate.
Rate of post-partum haemorrhagia | On the day of the delivery
  Rate of post-partum haemorrhagia above 500 mL, above 1000 mL, transfusion level and number of packed red blood cells transfused
Rate of uterine rupture | On the day of the delivery
  Number of patients with a uterine rupture
Rate of intra-uterine infections | On the day of the delivery
  Number of patients with intra-uterine infections (body temperature above 38°C measured twice within 30 minutes, associated to 2 criteria within the followings: foetal tachycardia above 160 beats per minute, pain of the uterus or painful uterus contractions ou spontaneous labour induction, or purulent amniotic fluid.
Rate of post-partum infections | One week after day of the delivery
  Number of patients with post-partum infections (body temperature above 38°C with antibiotic treatment, urinary tract infections, bacteriological endometritis)
Rate of neonatal asphyxia | On the day of the delivery
  Number of fetuses with neonatal asphyxia
Rate of hospitalization in Neonatal intensive care unit | Up to four days after the delivery
  Number of newborn babies hospitalized in Neonatal intensive care unit
Rate of proven bacteriological infections in newborn babies | Up to four days after the delivery
  Number of proven bacteriological infections in newborn babies
Rate of metrorrhagias while putting in place the dilatation balloon or the vaginal pad (dinoprostone) | On the day of the delivery
  Number of women who experienced metrorrhagias while putting in place the dilatation balloon or the vaginal pad (dinoprostone)
Pain level linked to the inflation of the dilatation balloon and requiring the partial deflation of the balloon | On the day of the delivery
  Measurement of Pain will be made using an Visual Analog Scale (VAS). The pain level will be linked to the inflation of the dilatation balloon and requiring the partial deflation of the balloon
Pain level recorded at different times of the labour induction | On the day of the delivery
  Measurement will be made using a Visual Analog Scale (VAS) and will be recorded at different times of the dilatation balloon or the dinoprostone vaginal pad set up
Assessment of the patient experience of the labour induction | Up to two weeks after the delivery
  Patient experience will be assessed using the W-DEQ (Wijma Delivery Expectancy/Experience Questionnaire)
Assessment of each strategy direct main costs | through study completion, an average of 3 years
  The costs of the treatment and duration of the hospitalization will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, MD PhD, Study Director — UH of Montpellier
Locations (2):
- France (2):
  - Montpellier University Hospital, Montpellier
  - Nimes University Hospital, Nîmes

IPD SHARING:
Plan to Share IPD: No